CLINICAL TRIAL: NCT00169507
Title: Phase III Multicentric Open Study to Evaluate Immunological Memory Induced by 3-dose Primary Vaccination Followed by Booster Dose of GSK Biologicals' 11-valent Conjugate Pneumococcal Vaccine Compared to Unprimed Subjects by Giving 1 Dose of Aventis Pasteur's Pneumo 23
Brief Title: Study of Immunological Memory Induced in Children by a Full 4 Dose Vaccination Schedule of 11 Valent Pneumococcal Conjugate Vaccine by Giving 1 Dose of Aventis Pasteur's 23-valent Pneumococcal Polysaccharide Vaccine (Pneumo 23)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104083
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Prophylaxis Pneumococcal Vaccine
MeSH Terms: interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: Pneumococcal (vaccine)

SUMMARY:
Evaluate the immunological memory induced by 4 doses of GSK Biologicals' 11valent pneumococcal vaccine; study antibody persistence 30 months after the 4 dose vaccination with GSK Biologicals' 11-valent pneumococcal vaccine in Undeca-Pn-010 study.

DETAILED DESCRIPTION:
Primed group: 50 subjects who previously received 4 doses of GSK Biologicals' 11Pn-PD vaccine will receive 1 dose of Pneumo 23 Unprimed group (Control): 50 subjects who received GSK Biologicals' Havrix™ vaccine will receive 1 dose of Pneumo 23

ELIGIBILITY:
Inclusion criteria: Male or female who participated in Undeca-Pn-010 study, were part of the blood subset and received 4 doses of GSK Biologicals' 11Pn-PD vaccine, or Havrix vaccine. Exclusion criteria: Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceeding the first dose of study vaccine, or planned use during the study period. Administration of any additional pneumococcal vaccine since study end of Undeca-Pn-010 (347414/010)

Ages: 31 Months to 57 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2005-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Antibody concentrations (ELISA) to pneumococcal serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F 10-15 days after the single dose of Aventis Pasteur's 23-valent pneumococcal polysaccharide vaccine (Pneumo 23).

SECONDARY OUTCOMES:
Before Pneumo 23 administration: Antibody concentrations (ELISA) to pneumococcal serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F & seropositivity (S+) status* (>= 0.05 µg/mL) * also measured 10-15 days after dose of Pneumo 23
Before and 10-15 days after dose of Pneumo 23: Antibody titers (opsono) to selected pneumococcal serotypes and S+ status (>= 8)
Occurrence of SAEs during study period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Slovakia (4):
  - GSK Investigational Site, Dubnica nad Váhom
  - GSK Investigational Site, Nová Dubnica
  - GSK Investigational Site, Považská Bystrica
  - GSK Investigational Site, Púchov

REFERENCES:
- [Derived] Schuerman L, Prymula R, Chrobok V, Dieussaert I, Poolman J. Kinetics of the immune response following pneumococcal PD conjugate vaccination. Vaccine. 2007 Mar 1;25(11):1953-61. doi: 10.1016/j.vaccine.2006.12.007. Epub 2006 Dec 26. PMID 17258358